CLINICAL TRIAL: NCT02256007
Title: Cognitive Motor Therapy Applications Using Videogame Platform
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible in inpatient setting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Blue Marble Rehab Inc (Industry)
Responsible Party: Principal Investigator, Pamela Roberts, Program Director, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00031722
Record Dates: First submitted 2014-09-28; First posted 2014-10-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Stroke
Keywords: Videogames; stroke
MeSH Terms: conditions — Stroke | interventions — Paper

STUDY DESIGN:
Intervention Model Description: Two treatment sessions during an inpatient rehabilitation stay. Part 1 is the screening (Montreal Cognitive Assessment and the Boston Diagnostic Aphasia Examination). Assessments will be given to make sure patient is eligible for the study. If eligible, will complete part 2-paper and pencil tasks and video game tests.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standardized Assessments (Active Comparator): Standardized Assessments (paper and pencil tests) to be given to each participant. The standardized assessments will be completed in paper and pencil format. These tests include:
  * Line Bisection Test
  * Patient Reported Outcomes
  * Trial Making A and B
  * Usability Questionnaire
  Interventions: Other: Paper and Pencil Assessments
- Videogame Assessments (Experimental): Videogame assessments will be performed by each participant using videogames. The videogame assessments will be performed using videogames on a tabletop platform with touchscreen which includes:
  * Line Crossing
  * Patient Reported Outcomes
  * Trial Making A & B-Asteroid Adventure Game
  * Usability Questionnaire
  Interventions: Other: Paper and Pencil Assessments

INTERVENTIONS:
Other: Paper and Pencil Assessments — Videogame Assessments

SUMMARY:
This study designs and develops an evidence-based game approach that will enhance the investigators understanding and usability of electronic tools to measure cognitive and sensorimotor abilities in an inpatient rehabilitation stroke population.

DETAILED DESCRIPTION:
The rehabilitation industry is the incipient stages of developing and using electronic based assessment and intervention tools. With the growing understanding of cognitive recovery following stroke, rehabilitation specialists are optimistic that appropriate rehabilitation interventions may optimize and enhance functional outcomes. The use of technology based assessments via video games may assist in a patient's cognitive recovery. Design and development of an evidence-based game approach will enhance the investigators understanding and usability of electronic tools to measure cognitive and sensorimotor abilities. There is no intervention only an assessment for usability.

ELIGIBILITY:
Inclusion Criteria:

* New onset stroke
* Ability to follow one-step commands

  * All participants must be admitted to the inpatient rehabilitation unit at Cedars-Sinai Medical Center
  * Scores needed for Participation in Study on the Complex Ideational Material-Short Form from the Boston Diagnostic Aphasia Examination and the Montreal Cognitive Assessment:
* Complex Ideational Material-Short Form from the Boston Diagnostic Aphasia Examination-Participants must obtain a total score of at least 5/6 item pairs to participate
* Montreal Cognitive Assessment-Participants must obtain a total score of 16 or greater and obtain a score of 6/6 on the orientation subtest
* In order to participate, participants must meet both of the above criteria

Exclusion Criteria:

* Patients who do not meet inclusion criteria as noted above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Usability Questionnaire | Session in which participant completes standardized assessments before the patient's discharge from inpatient rehabilitation (within 2 weeks)
  Participant will perform videogame assessments and standardized paper-pencil assessments and evaluate the utility of the touch screen tests compared to the traditional testing methods using the Usability Questionnaire. The focus will be on the Usability Questionnaire (not the video or paper assessments)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Roberts, PhD, Principal Investigator — Cedars-Sinai Medical Center; Jeffrey Wertheimer, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Pamela Roberts, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No subjects completed study

REFERENCES:
- [Background] King M, Hale L, Pekkari A, Persson M, Gregorsson M, Nilsson M. An affordable, computerised, table-based exercise system for stroke survivors. Disabil Rehabil Assist Technol. 2010 Jul;5(4):288-93. doi: 10.3109/17483101003718161. PMID 20302419
- [Background] Lewis GN, Rosie JA. Virtual reality games for movement rehabilitation in neurological conditions: how do we meet the needs and expectations of the users? Disabil Rehabil. 2012;34(22):1880-6. doi: 10.3109/09638288.2012.670036. Epub 2012 Apr 5. PMID 22480353
- [Background] Lewis GN, Woods C, Rosie JA, McPherson KM. Virtual reality games for rehabilitation of people with stroke: perspectives from the users. Disabil Rehabil Assist Technol. 2011;6(5):453-63. doi: 10.3109/17483107.2011.574310. Epub 2011 Apr 17. PMID 21495917